CLINICAL TRIAL: NCT07376928
Title: Multicenter Prospective Real-world Observational Study to Evaluate the Effectiveness of Phlebotonics, as Conservative Therapy in a Cohort of Patients With Symptomatic Hemorrhoidal Disease (HD) of I, II or III Goligher Grade
Acronym: VIVI2022/01
Status: Completed | Type: Observational
Sponsor: Italfarmaco (Industry)
Responsible Party: Sponsor
Other Study IDs: VIVI2022/01
Record Dates: First submitted 2026-01-13; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hemorrhoidal Disease
Keywords: Goligher grade I; Goligher grade II; Goligher grade III

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Phlebotonics
  Interventions: Drug: Phlebotonic

INTERVENTIONS:
Drug: Phlebotonic — Phlebotonics treatment will be used

SUMMARY:
Hemorrhoidal disease is one of the most common proctologic disease. This condition affects a large number of people in the world: the prevalence can vary from 4.4% in the general population to 36.4% in general practice [1]. It usually appears with symptoms and signs of bleeding, prolapse, soiling, itching, and pain. Bleeding is the most relevant and frequent symptom, reported by 56-81% of the patients; this sign is the most important reason for which most of patients are worried and they decide to be subjected to proctologic examination.

Medical and conservative management (life style changes, high-fiber diets, stool softeners, laxatives, and sitz baths are treatments chosen in hemorrhoidal disease from Goligher's I to III grade.

Hemorrhoidal disease (HD) has a significative incidence accounting for a large number of consultation per year and a large number of ambulatory or surgical treatments. Early symptoms are often treated tempirically with self prescription and OTC (over-the-counter) products with in spite of the value of different substances available.

In addition, symptoms such as tenesmus, mucus secretion or intense anal pain, if frequent and intense, significantly worsen the patient's quality of life and therefore require particular attention Phlebotonics are heterogeneous and widely investigated classes of drugs used to treat hemorrhoidal disease, with the aim to obtain strengthening of blood vessel walls, increasing venous tone, lymphatic drainage, normalizing capillary permeability, and anti-inflammatory effects.

Scientific production includes research on individual active ingredients but also on products that exploit the synergy of multiple active ingredients. Furthermore, the use of flavonoids is being analyzed both as an alternative to surgery, both in preparation and after the surgery itself.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent allowing data collection in accordance with local requirements;
* Males or females aged ≥ 18 years;
* Patients with symptomatic hemorrhoidal disease (HD) of I, II or III Goligher grade;
* Patients who are going to start treatment with phlebotonics, according to the clinical practice and according to the approved indications as described in the current version of the SmPC (Summary of Product Characteristics) approved in Italy. Patients are considered includible both in case never used phlebotonics or have stopped using phlebotonics for at least one month.

Exclusion Criteria:

* Presence of concomitant, severe systemic disorders;
* Hypersensitivity to the active ingredients of products under observation, or to one or more excipients present in the products under observation or known hypersensitivity to any other product containing the same active ingredients or excipients;
* History of Colorectal or anal cancer and/or radiotherapy; obstructive defecation syndrome; irritable bowel syndrome; inflammatory bowel disease; coagulation disorders; other proctologic diseases, such as anal abscess or fistula; anal fissure or acute hemorrhoidal thrombosis; and anticoagulant or anti-aggregant intake for another disease;
* Women who are known to be pregnant or breastfeeding;
* Current participation in another trial is not permitted unless it is a non-interventional study, and the sole purpose of the trial is for long-term follow up describing clinical features or survival data (registry).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic hemorrhoidal disease (HD) of I, II or III Goligher grade
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
The baseline characteristics of this italian real-world cohort | 36 months
  The primary endpoint has been evaluated using HDSS-Hemorrhoidal disease symptoms score by Rorvik.

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Piero Palagi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No